CLINICAL TRIAL: NCT02752763
Title: Comparison of Autologous Serum Versus Preservative Free Artificial Tear in Patients With Dry Eye Due to Systemic Isotretinoin Therapy
Brief Title: Comparison of Autologous Serum Versus Preservative Free Artificial Tear
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Niğde State Hospital (Other)
Responsible Party: Principal Investigator, Uğur Yılmaz, Opthalmologist M.D., Niğde State Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NSH 333
Record Dates: First submitted 2016-03-31; First posted 2016-04-27 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Dry Eye
Keywords: Dry eye; isotretinoin, AS; Autologous serum
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Ophthalmic Solutions; Polyvinyl Alcohol; Povidone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- preservative free artificial tear drop (Experimental): preservative free artificial tears drop is a drop group declaring different kind of active agent like hydroxypropyl methylcellulose, carboxymethyl cellulose etc commonly used in dry eye treatment. Preservative free artificial tear( carboxymethyl cellulose, hydroxypropyl methylcellulose) was used as four times one drop daily. In our study, we prescribed to patients preservative free artificial tears drop(hydroxypropyl methylcellulose or carboxymethyl cellulose) four times one drop daily.
  Interventions: Drug: Preservative free artificial tears(Tears naturale free, Refresh single dose eye drop)
- %40 Autologous serum(AS) (Experimental): peripheral venous blood (14-20 ml) that drawn from antecubital vein of patients to prepare Autologous Serum. Blood sample was left at room temperature over 2 hours for clotting. Serum was obtained after centrifugation at 4000 revolutions per minute (rpm) for 10 minutes at 4 °C using a Nuve NF1200R. Next, in a laminar flow cabinet under sterile conditions, approximately 10 mL of supernatant was collected and diluted to 40 % with isotonic saline solution. It is recommended for dry eye diseases, too. %40 diluted Autologous Serum used as four times one drop daily.
  Interventions: Drug: %40 diluted Autologous serum

INTERVENTIONS:
Drug: %40 diluted Autologous serum — Serum that obtained after centrifugation of blood sample
  Arms: %40 Autologous serum(AS)
Drug: Preservative free artificial tears(Tears naturale free, Refresh single dose eye drop) — Preservative free artificial tears is a group naming for drops commonly used for drye disease
  Other Names: Tears naturale free(hydroxypropyl methylcellulose); Refresh single dose(polyvinyl Alcohol + Povidone)
  Arms: preservative free artificial tear drop

SUMMARY:
Dry eye is a significant adverse effect of isotretinoin causing patients to use ophthalmic medications. For this reason, many patients using isotretinoin are referred to ophthalmology clinic because of discomfort symptoms. In the literature, there are studies suggesting superiority of Autologous serum drops regarding effects on ocular surface when compared to artificial tear. In addition, Autologous serum was also used in several corneal pathologies with successful outcomes. No data regarding use in the ocular adverse effects of isotretinoin was found in the literature; however, investigators think that it may be an effective alternative in the treatment of dry eye developed during isotretinoin use due to positive effects on ocular surface, epithelial regeneration and anti-inflammatory effect. Autologous serum can be a choice of ophthalmologists in routine practice by increasing number of comprehensive studies investigating effectiveness, safety and long-terms effects of Autologous serum therapy.In this study, it was aimed to investigate dry eye development in the patients receiving systemic retinoic acid therapy and to compare effectiveness of Autologous serum and Preservative free artificial tear in the patients with dry eye disease.

DETAILED DESCRIPTION:
This prospective, cross-sectional, double blind study was conducted by Ophthalmology Clinic on patients who have drye eye due to systemic isotretinoin treatment for several reasons in Niğde State Hospital between October, 2015 and March 2016. Patients determined as having drye eye during systemic isotretinoin treatment were included to our study. At baseline, 1.and 2. month of study, detailed ocular examination, best corrected visual acuity measurement, intraocular pressure measurement, Tear Break-Up time(TBUT)(5 µL of fluorescein sodium 2 % eye drops was used per each measurement using a pipette for standardization, and the mean value of two readings per patient was recorded) and Schirmer Test I (ST I) without topical anesthesia were performed. Effect on daily life was assessed by using Ocular Surface Disease Index (OSDI) score. TBUT<10 seconds, ST I <10 mm without local anesthesia, corneal and conjunctival staining was interpreted in favor of dry eye. In the follow-up period, investigators investigated the efficacy of autologous serum eye drops for the patients having dry eye illness during isotretinoin treatment. After informed consent, peripheral venous blood (14-20 ml) was drawn from antecubital vein of patients to prepare AS. Blood sample was left at room temperature over 2 hours for clotting. Serum was obtained after centrifugation at 4000 revolutions per minute (rpm) for 10 minutes at 4 °C using a centrifugal device(Nuve NF1200R). Next, in a laminar flow cabinet under sterile conditions, approximately 10 mL of supernatant was collected and diluted to 40 % with isotonic (0.9 % NaCl) saline solution and then 25 mL of preparation was aliquoted into 1.5-mL Eppendorf vials, each of which was wrapped with aluminum foil by the other specialist(Erkut Küçük) for protection against ultraviolet light (to prevent vitamin A degradation), and blinding the patients to the treatment. PFAT eye drops were also placed into different 1.5-ml Eppendorf vials and likewise wrapped with aluminum foil by the other specialist(Erkut Küçük) for blinding the patients. The droppers were also wrapped with aluminum foil for further blinding the patient while applying the eye drops. Patients were randomised via assigned laterality numbers and sealed regime envelopes by the other specialist(Erkut Küçük). Preservative-free isotonic saline was used for washout for 2 weeks prior to beginning of the study.

After the first treatment period (1 month) all patients underwent a 2-week washout period with isotonic saline (0.9 % NaCl) eye drops. Ten a new set of vials (AS or PFAT) was assigned to each patient by the other specialist(Erkut Küçük) for the second treatment period.

After the first 1-month treatment period, patients who had conventional PFAT treatment were switched to AS treatment and the patients who had AS treatment in the first 1-month treatment period were switched to conventional PFAT treat- ment in the second 1-month treatment period, according to the study's crossover nature. The examining ophthalmologist (Uğur Yılmaz) that performed tear function and ocular surface evaluations was blinded to the type of eye drops given to each patient. In addition, the patients were blinded to which treatment they were receiving.

Only the Other specialist (Erkut Küçük), who was not responsible for patient evaluation, knew which patient received which treatment during study periods. All patients were instructed to keep the vials (containing either AS or PFAT) in a refrigerator at 4 °C. All patients were advised to change the vial every other day during the treatment period. TBUT and ST I were administered by the same ophthalmologist (Uğur Yılmaz).

The study was approved Institutional Review Board of Erciyes University, Medicine School. The study was conducted in accordance to Helsinki Declaration. All patients gave written informed consent.

ELIGIBILITY:
Inclusion Criteria

• isotretinoin use for any reason

Exclusion Criteria:

* corneal pathologies such as dry eye illness before isotretinoin treatment
* previous cornea surgery, injury or keratitis
* active ocular infection
* meibomian gland dysfunction
* excessive allergic reaction that may be associated with dry eye
* glaucoma therapy use
* severe anemia
* previously use of PFAT or AS for any reason
* (Hb<10 g/dL) and elevated hepatic function tests requiring withdrawal of therapy

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in Schirmer Test I in Patients with Dry Eye due to isotretinoin use after autologous serum or preservative free artificial tears treatment | up to 3 Months monthly measurements were done
  Schirmer Test I is used for Dry Eye evaluation before and after autologous serum or preservative free artificial tears treatment. Schirmer test is used to measure tear secretion. Schirmer strips are used for this test. Wetting of the paper is recorded in millimeter
Change in Break up Time in Patients with Dry Eye due to isotretinoin use after autologous serum or preservative free artificial tears treatment | up to 3 Months monthly measurements were done
  fluorescein sodium eye drops was used for measurement of Break up Time. Value of Break up Time for per eye is recorded as seconds
Change in Ocular surface Disease Index in Patients with Dry Eye due to isotretinoin use after autologous serum or preservative free artificial tears treatment | up to 3 Months monthly measurements were done
  OSDI score is a reliable and feasible test which is commonly used for dry eye patients to grade either dry eye symptom severity and its effect on vision-related function. In this index, people are asked to indicate whether they experienced any of the symptoms or problems due to drye eye, if so, how often. Every question asked to patients is scored from one to four according to the frequency of symptoms. The scores were collected from all the questions.

CONTACTS AND LOCATIONS:
Overall Officials: Uğur Yılmaz, M.D., Study Chair — Niğde State Hospital
Locations (1):
- Niğde State Hospital, Niğde, Niğde Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Oner AF, Ferahbas A, Karakucuk S, Utas S, Karaman B, Kutlugun C et al. Ocular side effects associated with systemic isotretinoin. Cutan Ocul Toxicol. 2005;23:189-195.
- [Background] Egger SF, Huber-Spitzy V, Bohler K, Scholda C. [Isotretinoin administration in treatment of acne vulgaris. A prospective study of the kind and extent of ocular complications]. Ophthalmologe. 1995 Feb;92(1):17-20. German. PMID 7719068
- [Background] Tananuvat N, Daniell M, Sullivan LJ, Yi Q, McKelvie P, McCarty DJ, Taylor HR. Controlled study of the use of autologous serum in dry eye patients. Cornea. 2001 Nov;20(8):802-6. doi: 10.1097/00003226-200111000-00005. PMID 11685055
- [Background] Kojima T, Ishida R, Dogru M, Goto E, Matsumoto Y, Kaido M, Tsubota K. The effect of autologous serum eyedrops in the treatment of severe dry eye disease: a prospective randomized case-control study. Am J Ophthalmol. 2005 Feb;139(2):242-6. doi: 10.1016/j.ajo.2004.08.040. PMID 15733983
- [Background] Urzua CA, Vasquez DH, Huidobro A, Hernandez H, Alfaro J. Randomized double-blind clinical trial of autologous serum versus artificial tears in dry eye syndrome. Curr Eye Res. 2012 Aug;37(8):684-8. doi: 10.3109/02713683.2012.674609. Epub 2012 Jun 6. PMID 22670856